CLINICAL TRIAL: NCT03664310
Title: A Pilot Study and Randomized Controlled Trial of Transdiagnostic Sleep and Anxiety Treatment
Brief Title: Transdiagnostic Sleep and Anxiety Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018.23848
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSET Anxiety and Sleep Treatment (Experimental): The FSET Anxiety and Sleep Treatment (FAST) is a brief, 45-minute computerized intervention that can be accessed by any device connected to the Internet. The majority of the information is delivered via text. The program contains some interactive features such as quizzes, which direct participants to content, personalized to the individual user (for example screenshots, see Figure 2). FAST contains four modules: motivation, psychoeducation, behavioral tools, and behavior change.
  Interventions: Other: FSET Anxiety and Sleep Treatment
- Control (Active Comparator): The control condition is the Physical Health Education Treatment (PHET) used in several of our laboratory's prior studies (Schmidt, Capron, Raines, & Allan, 2014). PHET is also a 45-minute computerized intervention, including audio and visual features as well as comprehension quizzes.
  Interventions: Other: Control

INTERVENTIONS:
Other: FSET Anxiety and Sleep Treatment — Computerized anxiety and insomnia intervention.
  Arms: FSET Anxiety and Sleep Treatment
Other: Control — Physical health control
  Arms: Control

SUMMARY:
Background: Anxiety and insomnia disorders are two of the most common and costly mental health conditions. These disorders are frequently comorbid, but current treatment approaches do not target both. To streamline treatment for these commonly comorbid conditions, a novel, computerized intervention was developed targeting a transdiagnostic factor, safety aids, which are cognitive or behavioral strategies individuals use to cope with distress associated with anxiety or insomnia, that paradoxically exacerbate symptoms. A randomized controlled trial was conducted to determine the acceptability and efficacy of this newly developed intervention. Method: Young adults (N = 61) with elevated anxiety and insomnia symptoms were randomized to receive the anxiety-insomnia intervention or a computerized control condition focused on general physical health behaviors. After the intervention, participants were followed up at one week and one month and completed self-report measures.

ELIGIBILITY:
Inclusion Criteria:

* 1 SD above the mean in anxiety and insomnia symptoms
* Interest in improving anxiety and sleep

Exclusion Criteria:

* Participating in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-12 (Actual); Study Completion 2018-05-12 (Actual)

PRIMARY OUTCOMES:
Safety Aid Scale | Month 1
  safety aids. Total score (79-445). Higher score indicates worsened symptoms.

SECONDARY OUTCOMES:
Sleep Related Behavior Questionnaire | Month 1
  sleep safety aids. Total score (32-128). Higher scores indicate worse symptoms.
Penn State Worry Questionnaire | Month 1
  worry. Total score (16-80). Higher scores indicate worse symptoms.
Dimensional Obsessive Compulsive Scale | Month 1
  OC symptoms. Total score (0-80). Higher scores indicate worse symptoms.
Insomnia Severity Index | Month 1
  insomnia. Total score (0-28). Higher scores indicate worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States